CLINICAL TRIAL: NCT04112667
Title: Functionally Validated Structural Endpoints for Early AMD
Acronym: ALSTAR2
Status: Completed | Type: Observational
Sponsor: Cynthia Owsley (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Cynthia Owsley, Professor of Ophthalmology and Visual Sciences, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Other Study IDs: IRB-300003067; 1R01EY029595 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-06

CONDITIONS: Age-related Macular Degeneration; Aging
Keywords: vision; retina; dark adaptation; light sensitivity; spectral domain optical coherence tomography; quantitative autofluorescence; optical coherence tomography angiography
MeSH Terms: conditions — Macular Degeneration; Photophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum for DNA for genotyping. Serum for Biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Macular Health: >=60 years old with no macular disease
  Interventions: Other: Normal Macular Health
- Early Macular Degeneration: >=60 years old with early age-related macular degeneration
  Interventions: Other: Early Macular Degeneration
- Young Normals: 20-30 years old with normal macular health
  Interventions: Other: Young Normals

INTERVENTIONS:
Other: Normal Macular Health — This group of participants will have function assessed using rod- and cone-mediated tests (rod-mediated dark adaptation, 2 color dark adapted perimetry, cone-mediated perimetry, photopic and mesopic acuity, photopic and mesopic contrast sensitivity). Age-related macular degeneration status will be determined by multi-modal imaging.
  Groups: Normal Macular Health
Other: Early Macular Degeneration — This group of participants will have function assessed using rod- and cone-mediated tests (rod-mediated dark adaptation, 2 color dark adapted perimetry, cone-mediated perimetry, photopic and mesopic acuity, photopic and mesopic contrast sensitivity). Age-related macular degeneration status will be determined by multi-modal imaging.
  Groups: Early Macular Degeneration
Other: Young Normals — This group of participants will have function assessed using rod- and cone-mediated tests (rod-mediated dark adaptation, 2 color dark adapted perimetry, cone-mediated perimetry, photopic and mesopic acuity, photopic and mesopic contrast sensitivity). Age-related macular degeneration status will be determined by multi-modal imaging.
  Groups: Young Normals

SUMMARY:
Delayed rod-mediated dark adaptation (RMDA), or delayed recovery of vision in a dark environment, is a functional biomarker (i.e., risk factor) for early age-related macular degeneration (AMD). This research plan is designed to elucidate the structural (anatomical) basis of this visual deficit using cellular- and subcellular level imaging of the retina and its supporting tissues in living people. An accurate map and timeline of structure-function relationships in persons tested for night vision will result in functionally validated structural endpoints for early AMD trials, as well as define major biologic effects for development into future treatments.

DETAILED DESCRIPTION:
The Alabama Study on Early Age-Related Macular Degeneration 2 (ALSTAR2) is a prospective cohort study with baseline measurements that are repeated at follow-up 3 years later. The baseline and 3 year follow-up visits will each consist of 2 visits for a total of 4 visits.

Study assessments are listed below. All are collected at two visits at both baseline and follow-up for 4 visits total (blood collection for DNA analysis at baseline only). For some functional tests (photopic and mesonic acuity, photopic and mesonic contrast sensitivity), each eye will be tested separately. For other functional tests (dark-adapted two-color perimetry, light-adapted cone-mediate perimetry, rod-mediated dark adaptation), only one eye will be tested, which will be designated by the study eye. Tropicamide 1% and phenylephrine hydrochloride 2.5% are used to dilate pupils (diameter of ≥ 6 mm) as needed for specific parts of the protocol. After completing the baseline visits, participants will receive an annual phone call from the study coordinator so that contact information can be updated. Participants will receive an annual newsletter containing study related information (this will be submitted to the IRB for approval).

Study Assessments:

1. Rod-mediated dark adaptation (RMDA), the ability to recover light sensitivity after exposure to a bright light.
2. Dark-adapted two-color microperimetry, a measure of light sensitivity for lights of two different colors.
3. Photopic and mesopic acuity in central vision, as measured by letter charts..
4. Photopic and mesopic contrast sensitivity in central vision, as measured by letter charts..
5. Multimodal ocular imaging on both eyes, which consists of the following: color fundus photography, spectral domain optical coherence tomography (SDOCT), blue fundus autofluorescence (standard and quantitative), OCT-angiography (OCT-A).
6. Blood draw for the analysis of C-reactive protein, high-density lipoprotein, carotenoid level, DNA extraction, and examination of the presence of genetic risk associated with age-related macular degeneration (AMD).
7. Questionnaires: Demographics, medical co-morbidities, cognitive status screen, medication use, alcohol use, smoking, self-reported visual difficulty in the visual activities of daily living

The Young normal group will only complete:

1. Rod-mediated dark adaptation (RMDA), the ability to recover light sensitivity after exposure to a bright light.
2. Dark-adapted two-color microperimetry, a measure of light sensitivity for lights of two different colors.
3. . Photopic and mesopic acuity in central vision, as measured by letter charts..
4. Photopic and mesopic contrast sensitivity in central vision, as measured by letter charts..
5. Multimodal ocular imaging on both eyes, which consists of the following: color fundus photography, spectral domain optical coherence tomography (SDOCT), blue fundus autofluorescence (standard and quantitative),OCT-angiography (OCT-A).d and quantitative), OCT-angiography.

ELIGIBILITY:
Inclusion Criteria:

For those in Normal Macular Health or Early AMD: aged ≥ 60 years; either have normal macular health in both eyes at baseline or have early AMD in one eye For Young Normals: aged 20-30 years old; normal macular health in both eyes.

Exclusion Criteria:

Exclusion for those in normal macular health are:

* ANY EYE CONDITION OR DISEASE IN EITHER EITHER (OTHER THAN EARLY CATARACT) THAT CAN IMPAIR VISION INCLUDING:
* diabetic retinopathy
* glaucoma
* ocular hypertension
* history of retinal diseases (e.g., retinal vein occlusion, retinal degenerations)
* optic neuritis
* corneal disease
* previous ocular trauma or surgery
* REFRACTIVE ERROR >- 6 DIOPTERS
* NEUROLOGICAL CONDITIONS THAT CAN IMPAIR VISION OR JUDGEMENT INCLUDING:
* multiple sclerosis
* Parkinson disease
* stroke
* Alzheimer disease
* seizure disorders
* brain tumor
* traumatic brain injury
* PSYCHIATRIC DISORDERS THAT COULD IMPAIR THE ABILITY:
* to follow simple directions
* answer questions about health and functioning
* or to provide informed consent
* DIABETES
* ANY MEDICAL CONDITION THAT CAUSES SIGNIFICANT FRALITY OR IS BELIEVED TO BE TERMINAL.

Exclusion criteria for the early AMD group:

These are identical to those described above, except that it is acceptable for participants to have early AMD (AREDS 2-4) in one eye and be AREDS grade 1 or any stage of AMD in the fellow eye.

Exclusion for Young Normals:

* ANY EYE CONDITION OR DISEASE IN EITHER EYE (OTHER THAN EARLY CATARACT) THAT CAN IMPAIR VISION INCLUDING:
* diabetic retinopathy
* glaucoma
* ocular hypertension
* history of retinal diseases (e.g., retinal vein occlusion, retinal degenerations)
* optic neuritis, corneal disease
* previous ocular trauma or surgery
* RERACTIVE ERROR >=6 DIOPTORS
* NEUROLOGICAL CONDITIONS THAT CAN IMPAIR VISION OR JUDGEMENT INCLUDING:
* multiple sclerosis
* Parkinson disease
* stroke
* Alzheimer disease
* seizure disorders
* brain tumor
* traumatic brain injury
* PSYCHIATRIC DISORDERS THAT COULD IMPAIR THE ABILITY TO:
* follow simple directions
* answer questions about health and functioning
* or to provide informed consent
* DIABETES
* ANY MEDICAL CONDITION THAT CAUSES SIGNIFICANT FRAILTY OR IS BELIEVED TO BE TERMINAL.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: group 1 is >=60 years old with normal macular health group 2 is >=60 years old with early AMD group 3 is 20-30 years old are Young Normals
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Rod-mediated dark adaptation | Measured at baseline enrollment
  Time required to recover light sensitivity after exposure to bright light
Rod-mediated dark adaptation | Measured at 3 years after baseline enrollment
  Time required to recover light sensitivity after exposure to bright light
incident age-related macular degeneration (AMD) or progression of AMD using multimodal imaging | Measured at baseline enrollment
  development of AMD or progression of AMD at the 3 year follow up visit
incident age-related macular degeneration (AMD) or progression of AMD using multimodal imaging | Measured at 3 years after baseline enrollment
  development of AMD or progression of AMD at the 3 year follow up visit

SECONDARY OUTCOMES:
Light sensitivity as measured by microperimetry and perimetry | Measured at baseline enrollment
  Amount of light needed to detect a small target object
Light sensitivity as measured by microperimetry and perimetry | Measured at 3 years after baseline enrollment
  Amount of light needed to detect a small target object
Photopic and mesopic acuity | Measured at baseline enrollment
  Visual acuity under day time and twilight conditions
Photopic and mesopic acuity | Measured at 3 years after baseline enrollment
  Visual acuity under day time and twilight conditions
Photopic and mesopic contrast sensitivity | Measured at baseline enrollment
  Amount of contrast needed to recognize a letter under day time and twilight conditions
Photopic and mesopic contrast sensitivity | Measured at 3 years after baseline enrollment
  Amount of contrast needed to recognize a letter under day time and twilight conditions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Kar D, Corradetti G, Swain TA, Clark ME, McGwin G Jr, Owsley C, Sadda SR, Curcio CA. Choriocapillaris Impairment Is Associated With Delayed Rod-Mediated Dark Adaptation in Age-Related Macular Degeneration. Invest Ophthalmol Vis Sci. 2023 Sep 1;64(12):41. doi: 10.1167/iovs.64.12.41. PMID 37768273
- [Derived] Berlin A, Matney E, Jones SG, Clark ME, Swain TA, McGwin G Jr, Martindale RM, Sloan KR, Owsley C, Curcio CA. Discernibility of the Interdigitation Zone (IZ), a Potential Optical Coherence Tomography (OCT) Biomarker for Visual Dysfunction in Aging. Curr Eye Res. 2023 Nov;48(11):1050-1056. doi: 10.1080/02713683.2023.2240547. Epub 2023 Aug 4. PMID 37539829
- [Derived] McGwin G Jr, Kar D, Berlin A, Clark ME, Swain TA, Crosson JN, Sloan KR, Owsley C, Curcio CA. Macular and Plasma Xanthophylls Are Higher in Age-related Macular Degeneration than in Normal Aging: Alabama Study on Early Age-related Macular Degeneration 2 Baseline. Ophthalmol Sci. 2022 Dec 22;3(2):100263. doi: 10.1016/j.xops.2022.100263. eCollection 2023 Jun. PMID 36864830
- [Derived] Curcio CA, McGwin G Jr, Sadda SR, Hu Z, Clark ME, Sloan KR, Swain T, Crosson JN, Owsley C. Functionally validated imaging endpoints in the Alabama study on early age-related macular degeneration 2 (ALSTAR2): design and methods. BMC Ophthalmol. 2020 May 19;20(1):196. doi: 10.1186/s12886-020-01467-0. PMID 32429847